CLINICAL TRIAL: NCT04665505
Title: Resource Optimization in the Intensive Care Unit Setting: A Staff Education and Scheduling Pilot Study to Improve Treatment Decisions and Staff Satisfaction
Brief Title: Resource Optimization in the Intensive Care Unit Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Hopital Montfort (Other); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Kwadwo Kyeremanteng, Principal Investigator, Ottawa Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20200060-01
Record Dates: First submitted 2020-11-10; First posted 2020-12-11 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Burnout, Professional
Keywords: Resource Allocation; Personnel Staffing and Scheduling; Intensive Care Unit; Cost-Effectiveness; Burnout
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Single group data from the 6-month interventional period will be compared to data from the 3-month pre and post interventional periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICU Staff (Experimental): The study group is composed of ICU care providers at the Ottawa Hospital Civic campus and the Montfort Hospital, including intensivists, fellows, nurses and allied health professionals. The study site participant breakdown is approximately 58 TOH staff respondents and 15 Montfort respondents.
  Interventions: Behavioral: Educational Workshop; Behavioral: Optimizing Staff Scheduling

INTERVENTIONS:
Behavioral: Educational Workshop — The intervention consists of providing educational content for all ICU care providers concerning building staff knowledge surrounding methods to facilitate cost-effective and evidence-based decision-making about patient care (including tests, treatments, and procedures). The first intervention is an educational workshop to increase staffs' awareness of the current Choosing Wisely Canada Critical Care strategies and recommendations to facilitate cost-effective and evidence-based decision-making about patient care (including tests, treatments, and procedures).
Behavioral: Optimizing Staff Scheduling — This initiative will focus solely on the nurse subgroup and concerns schedule optimization to ensure the presence of the appropriate number of nurses per shift, thereby reducing stress, burnout and limiting the need for overtime.

SUMMARY:
The purpose of the study is to facilitate cost-effective, high quality care within the the ICUs of two Ottawa teaching hospitals through educational workshops and nurse scheduling optimization.

DETAILED DESCRIPTION:
This intervention pilot study has been developed for Intensive Care Unit (ICU) physicians and nurses by the Resource Optimization Network (RON) for implementation in The Ottawa Hospital (TOH) Civic Campus and the Montfort Hospital. The intervention targets ICU staff and is designed to reduce overall costs associated with ICU health care service delivery and improve staff satisfaction through reducing stress and associated burnout without sacrificing quality of care and patient outcomes. The intervention involves two components that (a) build ICU staffs' (i.e. physicians and nurses) knowledge to facilitate cost-effective and evidence-based decision making about patient care (including tests, treatments, and procedures); and (b) optimize nurse scheduling to ensure the presence of the appropriate number of nurses per shift, thereby reducing stress, burnout and limiting the need for overtime. To evaluate the impact of the intervention, a pre/post-intervention design will be employed, with a 3-month pre-intervention period, followed by a 6-month intervention period and a 3-month post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Employees aged 18 year and older who provide direct patient care in the ICU at the Civic Campus of the Ottawa Hospital or the Montfort Hospital as physicians, nurses, or allied health professionals (e.g., respiratory therapists, occupational therapists).

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
ICU Costs | 12 months
  Case costing will be used to determine the costs associated with ICU care during the study period, including: a) ICU total costs; b) ICU direct costs (i.e., all expenses to the hospital with fee codes linked to patient chart); c) ICU indirect costs (i.e., any overhead operational fees associated with service provided to patient); d) ICU cost/patient.
ICU Quality Metric 1: Ventilator Associated Pneumonia | 12 months
  This outcome will be included to evaluate the quality of ICU patient care during the study period. The number of patients who develop ventilator associated pneumonia will be collected from the TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Quality Metric 2: Central Line Infections | 12 Months
  This outcome will be included to evaluate the quality of ICU patient care during the study period. The number of patients who develop central line infections will be collected from the TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Quality Metric 3: C. difficile | 12 Months
  This outcome will be included to evaluate the quality of ICU patient care during the study period. The number of patients who develop C. difficile infections will be collected from the TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Quality Metric 4: Early Mobilization | 12 Months
  This outcome will be included to evaluate the quality of ICU patient care during the study period. The number of patients who receive early mobilization will be collected from the TOH Data Warehouse and Montfort's Department of Archives and Decision Support.

SECONDARY OUTCOMES:
ICU Patient Outcomes 1: Length of Stay | 12 Months
  Metrics for evaluation concerning patient outcomes include measurement of length of stay within the ICU in days, or LOS. Patient data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Patient Outcomes 2: Patient Deaths | 12 Months
  Metrics for evaluation concerning patient outcomes include measurement of the number of patients who die within the ICU. Patient data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Patient Outcomes 3: Perceived Quality of Care | 12 Months
  Metrics for evaluation concerning patient outcomes include measurement of the quality of care perceived by patients and their families. Data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Medical Procedures 1: Albumin Use | 12 Months
  Metrics for evaluation concerning ICU medical procedures specifically targeted in the educational intervention component include the rate of albumin used per ICU admission (bags of albumin used/admission). Patient data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Medical Procedures 2: Mechanical Ventilation | 12 Months
  Metrics for evaluation concerning ICU medical procedures specifically targeted in the educational intervention component include the number of patients mechanically ventilated, and the duration of their ventilation in days. Patient data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Medical Procedures 3: Chest Radiographs | 12 Months
  Metrics for evaluation concerning ICU medical procedures specifically targeted in the educational intervention component include the number of ICU patient chest radiographs completed per day. Patient data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
ICU Medical Procedures 4: Red Blood Cell Transfusions | 12 Months
  Metrics for evaluation concerning ICU medical procedures specifically targeted in the educational intervention component include the rate of red blood cell transfusions per admission. The amount of red blood cell transfusions administered (measured in bags/admission) will be monitored throughout ICU admission. Patient data used for this analysis will be collected from TOH Data Warehouse and Montfort's Department of Archives and Decision Support.
Rate of ICU Staff Absenteeism | 12 Months
  We will collect data on ICU full-time staff absenteeism during the study period from the Data Warehouse and Montfort Archives.
Stakeholder perceptions | 12 Months
  8-15 ICU stakeholder staff with special knowledge of ICU activities will be recruited for post-interventional interviews. The semi-structured interviews will be conducted by trained research staff and will use the Post-Intervention Semi-Structured Interview Guide to assess the stakeholders' perceptions of intervention outcomes. Stakeholders will be asked open-ended questions about their knowledge of the interventions implemented during the study period, their perceptions of the outcomes of these interventions, and any perceived changes in ICU care delivery in time period that corresponds to the post-intervention phase of the study. The interview will last approximately 30 minutes and will be digitally recorded and transcribed. Specific topics of discussion include introduction, participant's definition/perception of their field, quality of care, team morale/staff satisfaction and final thoughts/comments.
Staff Demographic Variable Collection 1 | 12 months
  A 15-20 minute self-administered online questionnaire will be used to obtain demographic information. It will include 9 questions, 6 of which are qualitative such as ICU role, part time or full time status, types of shifts worked, age group, gender identity (optional), and staff turnover.
  The 3 quantitative questions are measured from 0-5, where 0 is strongly disagree/very dissatisfied and 5 is strongly agree/very satisfied.
  Satisfaction relates to both job satisfaction and perceptions on whether staffing is efficient and promotes quality of care.
  Perceptions on quality of care will be measured based on agreement with the statement "there are adequate support services to allow sufficient patient interactions".
  Team morale has 3 sub questions: whether ICU physicians, nurses and allied health professional have good working relations, whether supervisory staff is supportive of ICU staff and whether there is sufficient teamwork between health care professionals.
Staff Demographic Variable Collection 2 | 12 months
  The Education Evaluation Survey will be administered at the end of the workshop and emailed the day after to obtain post-intervention data. Participants will identify their job position and any prior knowledge relating to test/treatment/procedure misuse in Canadian hospitals. They will detail their comfort prior to the workshop in engaging in conversations with patients about reducing unnecessary standard tests/treatments.
  Questions 4-8 can be answered by agree, neutral, disagree, don't know/non-applicable.
  I enjoyed the workshop, topic and lecture. I enjoyed the discussion among my peers. I have an increased awareness of what standard tests, treatments and procedures may be unnecessary or even harmful to my patients. I feel more comfortable about sharing knowledge with my peers and patients about what standard tests, treatments and procedures may be unnecessary or even harmful to my patients. I am more likely to engage in reflexive practices related to my healthcare practice.
Staff Stress Levels and Burnout 1 | 12 months
  The short self-administered online questionnaire will evaluate ICU staff stress and burnout, as well as demographic variables discussed above. It will contain questions from the Perceived Stress Scale (PSS).
  The PSS consists of 10 questions, answered on a scale of 0-4 depending on the frequency of which the behavior is observed, with 0 indicating "never" and 4 indicating "very often". Overall, a score of 0 indicates low stress, while a score of 40 indicates an individual with high perceived stress levels.
Staff Stress Levels and Burnout 2 | 12 months
  The short self-administered online questionnaire will evaluate ICU staff stress and burnout, as well as demographic variables discussed above. It will contain questions from the Maslach Burnout Inventory (MBI).
  The MBI is a 22 question survey which evaluates 3 subscales; emotional exhaustion, depersonalization and reduced personal accomplishment. Each question is rated from 1 to 5, where 1 is strongly disagree and 5 is strongly agree. A high score on the emotional exhaustion subscale (27+) coupled with a high score on the depersonalization scale (10+) indicates that the individual may be experiencing 1+ symptoms of burnout.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT04665505/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT04665505/ICF_001.pdf